CLINICAL TRIAL: NCT00966173
Title: An International, Multicenter, Prospective, Non-controlled, Non-randomised, Clinical Study to Collect Impedance Data of Potentially Malignant Pigmented Nevi and Histological Diagnoses
Brief Title: International Melanoma Algorithm Training Study - IMATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciBase AB (Other)
Responsible Party: Anders Lundqvist, CEO, SciBase AB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6001
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SciBase III Electrical Impedance Spectrometer — Following enrollment, patients will undergo measurements with SciBase III Electrical Impedance Spectrometer. Electrical impedance of the skin will be measured with a microinvasive spiked probe.

SUMMARY:
This is an international, multicenter, prospective, non controlled, non randomized, clinical study to collect electrical impedance data of potentially malignant pigmented nevi and histological diagnoses (International Melanoma Algorithm Training Study [IMATS]). The study objective is to collect data for training and optimization of an algorithm that can classify skin lesions using electrical impedance, i.e., to identify malignant melanomas.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any ethnic group
* Lesion located on normal healthy skin
* Maximum number of eight lesions per patient
* etc.

Exclusion Criteria:

* Lesion under finger and toe nails
* Lesion located on eczema, psoriasis areas or similar
* Lesion located on scars
* etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2005-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Outcome measure not applicable. This is an algorithm training study. | Q1 2010

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Dpt. of Dermatology, Gothenburg, Sweden